CLINICAL TRIAL: NCT01404949
Title: Phase II Study of Combined Tretinoin and Arsenic Trioxide for Patients With Newly Diagnosed Acute Promyelocytic Leukemia Followed by Risk-Adapted Postremission Therapy
Brief Title: Combined Tretinoin and Arsenic Trioxide for Patients With Newly Diagnosed Acute Promyelocytic Leukemia Followed by Risk-Adapted Postremission Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Northwestern University (Other); New York Presbyterian Hospital (Other); University of Southern California (Other); Princess Margaret Hospital, Canada (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-040
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-02

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Tretinoin; all-trans retinoic acid; ATRA; Vesanoid; Arsenic Trioxide; ATO; Trisenox; 11-040
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Tretinoin; Arsenic Trioxide

ARMS (1):
- Tretinoin and Arsenic Trioxide (Experimental): This is a multicenter, phase II trial to study the efficacy of combined tretinoin and ATO in the treatment of newly diagnosed APL in an effort to reduce or eliminate the amount of standard chemotherapy required for long-term remission.
  Interventions: Drug: Tretinoin and Arsenic Trioxide

INTERVENTIONS:
Drug: Tretinoin and Arsenic Trioxide — See Detailed Description

SUMMARY:
The purpose of this study is to find what effects, good and/or bad, treatment with two drugs has on leukemia. The first medicine is tretinoin (also called all-trans retinoic acid, ATRA, or Vesanoid). It is an approved medicine that causes the leukemia cells in APL to mature. It is related to vitamin A. The second is arsenic trioxide (Trisenox). It is an approved medicine for APL that comes back after earlier treatment.

APL is most often treated with tretinoin and standard chemotherapy drugs. These chemotherapy drugs can cause infection and bleeding. They can also damage the heart and normal bone marrow cells. This can lead to a second leukemia years later.

In this study, the investigators are using tretinoin and arsenic trioxide together. Both drugs work to treat APL. They have been used together in only a limited number of people. The investigators want to use these drugs together to reduce the amount of standard chemotherapy and decrease side effects. The patient will receive standard chemotherapy with a drug called idarubicin only if they have a higher chance of the leukemia coming back or a higher risk of side effects.

DETAILED DESCRIPTION:
Induction will consist of tretinoin 45 mg/m2 po daily (rounded up to the nearest 10mg) in two divided doses (25 mg/m2 in patients <20 years of age) for 35 days and ATO 0.15 mg/kg IV daily for 35 doses given 5-7 days per week. The drugs will then be discontinued, and the patient will be followed until a clinical complete remission is achieved. Idarubicin 12 mg/m2 IV for 4 doses will be added during induction on day 2 if the presenting WBC is >10,000/μl, or if the WBC increases to 5,000/μl on day 5, 10,000/μl on day 10, or 15,000/μl on day 15, because of the increased risk of the APL differentiation syndrome and relapse in these patients. Dexamethasone 10 mg twice daily with be given on days 1-14 of induction as prophylaxis for the APL differentiation syndrome. All patients will then receive four courses of consolidation with tretinoin 45 mg/m2 po daily (rounded up to the nearest 10mg) (25 mg/m2 in patients <20 years of age) for 15 days and ATO 0.15 mg/kg IV for 25 doses.

Patients with high-risk disease or who received Idarubicin during Induction may receive intrathecal cytarabine as CNS prophylaxis given by the treating physician during consolidation, at the discretion of the site PI. High-risk patients will also receive maintenance therapy with additional courses of tretinoin and ATO every 3 months for 2 years. Each maintenance course will consist of tretinoin 45 mg/m2 po daily (25 mg/m2 in patients <20 years of age) for 15 days and ATO 0.15 mg/kg IV for 10 doses. Disease status will be monitored with serial analyses of peripheral blood samples using RT-PCR for PML-RARα mRNA. Patients will be followed until relapse, death, loss to follow-up, or removal from study.

Induction therapy can be given as an inpatient or outpatient. Consolidation and maintenance treatments will be given as an outpatient. Consolidation may also be given at the patient's local institution. Intrathecal cytarabine treatments will be administered as an outpatient.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with a morphologic diagnosis of APL, confirmed by demonstration of t(15;17) using conventional cytogenetics OR florescence in situ hybridization (FISH), OR a positive RT-PCR assay for PML-RAR at the subject's local institution.
* Age ≥18 years. Karnofsky performance status of ≥ 60%.
* Adequate renal function as demonstrated by a serum creatinine ≤ 2.0 mg/dl or a creatinine clearance of > 60 ml/min.
* Adequate hepatic function as demonstrated by a bilirubin < 2.0 mg/dl (unless attributable to Gilbert's disease) and an alkaline phosphatase, AST, and ALT ≤ 2.5 times the upper limit of normal.
* Normal cardiac function as demonstrated by a left ventricular ejection fraction ≥ 50% on echocardiogram or MUGA scan.
* QTc ≤ 500 msec on baseline ECG.
* Negative serum pregnancy test in women of childbearing potential.
* Ability to swallow oral medication.
* Men and women of child-bearing potential must be willing to practice an effective method of birth control during treatment and at least 4 months after treatment is finished.
* Patients with central nervous system involvement by APL are eligible and may receive concomitant treatment with radiation therapy and/or intrathecal chemotherapy in accordance with standard medical practice.

Exclusion Criteria:

* Previous treatment for APL, except tretinoin, which may be given for up to 7 days prior to study entry.
* Active serious infections not controlled by antibiotics.
* Pregnant women or women who are breast-feeding.
* Concurrent active malignancy requiring immediate therapy.
* Clinically significant cardiac disease (NY Heart Association Class III or IV), including chronic arrhythmias, or pulmonary disease.
* Other serious or life-threatening conditions deemed unacceptable by the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-07; Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (12):
- United States (11):
  - University of Southern California, Los Angeles, California
  - Northwestern University, Evanston, Illinois
  - National Heart, Lung, and Blood Institute (NIH), Bethesda, Maryland
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital-Weill Medical College of Cornell University, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Cleveland Clinic, Cleveland, Ohio
- Princess Margaret Hospital/Ontario Cancer Institute, Toronto, Ontario, Canada

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tretinoin and Arsenic Trioxide
Started | 17
Completed | 16
Not Completed | 1
Not completed — Not Treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tretinoin and Arsenic Trioxide
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 54 [27 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Rate of Molecular Remission
Description: after induction with combined tretinoin and ATO (along with idarubicin in patients with high-risk disease or who develop leukocytosis) in APL.
Time Frame: 4 years
Population: Data were not collected
Arm/Group | Tretinoin and Arsenic Trioxide
Number analyzed (Participants) | 0

2. Secondary Outcome: Participants Who Experienced a Complete Remission
Description: after induction with tretinoin and ATO (with idarubicin in patients with high-risk disease or who develop leukocytosis).
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Tretinoin and Arsenic Trioxide
Number analyzed (Participants) | 16
Participants | 16

3. Secondary Outcome: To Determine the Proportion of Patients in Molecular Remission
Description: after each course of postremission therapy.
Time Frame: 4 years
Population: Data were not collected
Arm/Group | Tretinoin and Arsenic Trioxide
Number analyzed (Participants) | 0

4. Secondary Outcome: To Determine the Disease-free and Event-free Survival of Patients
Description: treated with this program.
Time Frame: 4 years
Population: Data were not collected
Arm/Group | Tretinoin and Arsenic Trioxide
Number analyzed (Participants) | 0

5. Secondary Outcome: To Determine the Toxicity of This Treatment Program
Description: including the early death rate (within 30 days), the incidence of APL differentiation syndrome, the number and length of hospitalizations, the incidence of secondary myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML), and the effects of treatment on left ventricular ejection fraction (LVEF) Frequencies of toxicities based on the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 will be tabulated.
Time Frame: 4 years
Population: Data were not collected
Arm/Group | Tretinoin and Arsenic Trioxide
Number analyzed (Participants) | 0

6. Secondary Outcome: To Characterize the Differentiation of APL Cells During Treatment
Description: with combined tretinoin and ATO using serial immunophenotyping studies of peripheral blood
Time Frame: 4 years
Population: Data were not collected
Arm/Group | Tretinoin and Arsenic Trioxide
Number analyzed (Participants) | 0

7. Secondary Outcome: Explore the in Vivo Induction of Telomerase-dependent Cell Death
Description: by ATRA (Tretinoin) and ATO (Arsenic Trioxide). Bone marrow samples will be analyzed at baseline and at the time of clinical CR for telomerase activity, telomere length and TERT expression
Time Frame: 4 years
Population: Data were not collected
Arm/Group | Tretinoin and Arsenic Trioxide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Tretinoin and Arsenic Trioxide
All-Cause Mortality (participants affected / at risk) | 2/17
Serious Adverse Events (participants affected / at risk) | 7/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tretinoin and Arsenic Trioxide (N=17)
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Delirium (Psychiatric disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Skin infection (Infections and infestations) | 1
Thromboembolic event (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tretinoin and Arsenic Trioxide (N=17)
Dry skin (Skin and subcutaneous tissue disorders) | 4
Fatigue (General disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 3
Eye disorders - Other, specify (Eye disorders) | 3
Headache (Nervous system disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Alkaline phosphatase increased (Investigations) | 2
Anemia (Blood and lymphatic system disorders) | 2
Aspartate aminotransferase increased (Investigations) | 2
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 2
Lymphocyte count decreased (Investigations) | 2
Nail ridging (Skin and subcutaneous tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Skin & subcutaneous tissue disordered Others, spec (Skin and subcutaneous tissue disorders) | 2
Weight loss (Investigations) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Alanine aminotransferase increase (Investigations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Blood bilirubin increased (Investigations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Cholesterol high (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Depression (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 1
Dry eye (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema limbs (General disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Gen disorders & admin site conditions Other, spec (General disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Hypertension (Vascular disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Insomnia (Psychiatric disorders) | 1
Investigation - Other, specify (Investigations) | 1
Lethargy (Nervous system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Myocarditis (Cardiac disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Platelet count decreased (Investigations) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1
Superficial thrombophlebitis (Vascular disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
White blood cell decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT01404949/Prot_SAP_000.pdf